CLINICAL TRIAL: NCT02981914
Title: Pilot Study of Pembrolizumab Treatment for Disease Relapse After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1195
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Classical Hodgkin Lymphoma; B-cell Non-Hodgkin Lymphoma; Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Classical Hodgkin Lymphoma; B-cell Non-Hodgkin Lymphoma; Acute Myeloid Leukemia; Myelodysplastic Syndromes; pembrolizumab
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be administered at a fixed dose of 200 mg IV every 3 weeks. Treatment will be administered for up to 24 months, provided that neither disease progression, nor development of a dose-limiting toxicity (DLT), has occurred.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered at a fixed dose of 200 mg IV every 3 weeks for a max of 24 months, so long as there is no disease progression.

SUMMARY:
This pilot study has been designed to investigate the safety of pembrolizumab treatment for disease relapse following allogeneic stem cell transplant (alloSCT). Pembrolizumab will be administered at a fixed dose of 200 mg IV every 3 weeks. Approximately 12-26 patients with relapsed MDS, AML, or mature B cell (B-NHL, cHL) malignancies that have relapsed following alloSCT will be enrolled on this trial. Pembrolizumab treatment will be administered for up to 24 months, provided that neither disease progression, nor development of a dose-limiting toxicity (DLT), has occurred. Adverse events will be monitored every three weeks throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. This trial will be conducted in accordance with Good Clinical Practices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with AML, MDS or mature B cell lymphomas that have relapsed following matched-related donor (MRD) or matched unrelated donor (MUD) (HLA-A -B -C -DR -DQ) alloSCT are eligible for enrollment

  1. Signed written informed consent

     1. Subjects must have signed and dated an IRB-approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
     2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
  2. Target population

     1. Subjects must be ≥ 18 years of age.
     2. Subjects must have an ECOG performance status of 0-1 (Appendix).
     3. Subjects have undergone alloSCT > 90 days prior to enrollment from a matched-related donor (MRD), matched-unrelated donor (MUD), cord blood donor, or haplo-identical and cord blood donor.
     4. There must be histological confirmation of relapse after alloSCT of any of the following diseases: any mature B cell lymphoma (cHL or NHL), AML or MDS.
     5. Subjects must be off of all immunosuppressive medications for a minimum of 2 weeks with the exception of physiologic doses of corticosteroids.
     6. Subjects with B cell lymphoma must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 2 dimensions with CT scan. Minimum measurement must be > 15 mm in the longest diameter and > 10 mm in the short axis.
     7. Subjects must not have had any prior investigational agents or devices within 4 weeks of beginning study drug
     8. Subjects must have no prior history of VOD
     9. Subjects must demonstrate adequate organ function as defined below. All screening labs should be performed within 10 days of treatment initiation.

        Hematological Absolute neutrophil count (ANC) ≥ 500 /mcL Platelets ≥ 20,000 /mcL Hemoglobin ≥ 8 g/dL (RBC transfusions are OK)

        Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X upper limit of normal (ULN) or
        * 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

        Hepatic Serum total bilirubin ≤ 1.5 X ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5X ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN Albumin ≥ 2.0 mg/dL

        Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy, in which case, the PT/INR should be within therapeutic range for intended use. Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy, in which case, the PTT should be within therapeutic range for intended use.

        *Creatinine clearance should be calculated per institutional standard.
     10. Female subjects of childbearing potential should have a negative urine or serum pregnancy test (β-hCG) within 72 hours prior to receiving the first dose of study medication.
     11. Female subjects with childbearing potential should be willing to use 2 methods of contraception, be surgically sterile, or abstain from heterosexual activity throughout the course of the study, until 120 days after the final dose of study medication. Subjects with childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Abstinence is acceptable if this is the established and preferred contraceptive method for the subject.
     12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study medication until 120 days after the final dose of study medicine. Abstinence is acceptable if this is the established and preferred contraceptive method for the subject.

Exclusion Criteria:

* 1. Target disease exclusions

  1. Subjects must not have known central nervous system involvement by disease (parenchymal, meningeal or cerebrospinal fluid) 2. Medical history, concurrent diseases, and prior treatments

  <!-- -->

  1. Subjects must not have a history of any positive test for hepatitis B or hepatitis C indicating active disease or previous exposure.
  2. Subjects must not have a history of human immunodeficiency virus (HIV) infection.
  3. Subjects must not be receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks prior to the first dose of study medication. The use of physiologic doses of corticosteroids is acceptable.
  4. Subjects must not be concurrently receiving disease-modifying therapy in another therapeutic investigational study.
  5. Subjects must not have received a prior monoclonal antibody within 4 weeks prior to the first dose of study medication, and must have recovered (≤ grade 1) from adverse events related to any anti-cancer agent administered > 4 weeks previous to the first dose of study medication.
  6. Subjects must not have received chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study medication, and must have recovered (≤ grade 1) from adverse events related to a previously administered agent.
  7. Subjects must not have received a donor lymphocyte infusion (DLI) within 8 weeks prior to the first dose of study medication.
  8. Subjects must not have a history of severe (grade 3-4) acute GVHD, and/or current > grade 1 acute GHVD. Subjects must not have a history of chronic GVHD (whether limited or extensive stage).
  9. Subjects must not have autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  10. Subjects must not have a known history of congestive heart failure, unstable angina pectoris, or cardiac arrhythmia (with the exception of chronic and rate-controlled atrial fibrillation).
  11. Subjects must not have a history of other serious underlying medical or psychiatric condition that, in the opinion of the investigator, would impair the ability to receive, tolerate and or comply with the planned treatment and follow-up.
  12. Subjects must not have a history of a known secondary primary malignancy that is not in remission and/or that requires active therapy. Exceptions include non-melanoma skin cancers and in situ cervical cancer that has undergone curative-intent local therapy.
  13. Subjects must not have a known active infection requiring intravenous antibiotic therapy.
  14. Subjects must not have a history of (non-infectious) pneumonitis that required steroid treatment, evidence of interstitial lung disease, or active, non-infectious pneumonitis. Subjects must not have active, non-infectious colitis.
  15. Subjects must not be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the final dose of study medication.
  16. Subjects must not have received a live vaccine within 30 days prior to the first dose of study medication.
  17. Subjects must not be or have an immediate family member (spouse, parent, legal guardian, sibling or child) who is an investigational site sponsor or staff directly involved with the trial, unless IRB approval is granted previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Kline, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Godfrey J, Liu H, Yu J, Tallarico M, Curran E, Artz A, Riedell PA, Stock W, Karrison T, Fitzpatrick C, Venkataraman G, Cooper A, Smith SM, Bishop MR, Kline J. Pembrolizumab for the treatment of disease relapse after allogeneic hematopoietic stem cell transplantation. Blood Adv. 2023 Mar 28;7(6):963-970. doi: 10.1182/bloodadvances.2022008403. PMID 35973200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 50.7 [26 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities (DLTs)
Description: A DLT is defined as the development of grade 3 or 4 acute GVHD (defined by the Gluckenberg scale), graft rejection, the development of any unexpected grade > 2 toxicity felt to be related to pembrolizumab, or the development of > grade 2 dysfunction of a vital organ felt to be secondary to an immune-related adverse event within 90 days following the initiation of pembrolizumab treatment.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
Participants | 3

2. Secondary Outcome: Time Between Initial Response and Subsequent Disease Progression or Relapse
Description: To determine the duration of response (DOR) of patients treated with pembrolizumab in the setting of relapsed myeloid malignancies and mature B cell lymphomas following alloSCT.
Time Frame: From date of response until the date of first documented progression or relapse, whichever came first, assessed up to 12 months
Population: Note: one patient censored at 54 days, second patient had disease progression at 364 days. Per the area under the Kaplan-Meier curve, the mean would be estimated as 364 days. However this estimate is unreliable given that it is based on only one censored observation and one event. The censored observation has been omitted in the full range below, as "54+" is rejected as a valid entry.
Measure: Mean (Full Range); unit: days
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 2
days | 364 [364 to 364]

3. Secondary Outcome: Objective Response Rate
Description: For B cell lymphoma patients, partial and complete responses will be defined according to the International Working Group criteria. For MDS patients, partial and complete responses (including cytogenetic responses) will be defined according to the International Working Group criteria. Lastly, for AML patients, complete (including CR, CRp, CRi), and partial responses will be defined according to the European Leukemia Net response criteria.
Time Frame: 24 months
Population: The trial enrolled 8 AML patients, 3 lymphoma patients, and 1 MDS patient. Both responders were lymphoma patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Time Between the Start of Therapy to Death From Any Cause.
Description: Survival time in days, patients alive as of last follow-up were censored
Time Frame: From start date of therapy to the date of death from any cause, whichever may come first, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
days | 285 [21 to NA] — NA = Upper confidence limit cannot be estimated due to insufficient number of participants with events

5. Other Pre Specified Outcome: Effect on Restoring Donor Chimerism
Description: To determine the effect of pembrolizumab on restoring donor chimerism in patients with relapsed myeloid malignancies and mature B cell lymphomas following alloSCT.
Time Frame: 24 months
Population: Data were not collected.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Effect of Pembrolizumab on the Numbers and Activations Status of Peripheral Blood T Cells
Time Frame: 24 months
Population: Data were not collected.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Compare PD-L1 Expression on Malignant Cells at Initial Diagnosis and at Disease Relapse Following alloSCT
Time Frame: 24 months
Population: Data were not collected.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Effect of Pembrolizumab on the T Cell Receptor (TCR) Repertoire in the Peripheral Blood, and Where Available, Tumor Environment, Following alloSCT
Time Frame: 24 months
Population: Data were not collected.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 7/12
Serious Adverse Events (participants affected / at risk) | 7/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=12)
Secondary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelet count decreased (Investigations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Infections and infestations) | 1
Hemolytic anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=12)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Autoimmune hemolytic anemia (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Coronavirus PNA (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Crackles (bilateral) (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Diverticulitis (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Ecchymoses (Injury, poisoning and procedural complications) | 1
Edema (General disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Enterocolitis infectious (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 7
Gum bleeding (General disorders) | 1
Headache (Nervous system disorders) | 3
Hematuria (Renal and urinary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
High FT4 (Investigations) | 1
Hypertension (Vascular disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 4
Hypothyroidism (Endocrine disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Low TSH (Investigations) | 1
Mild scleral icterus (Hepatobiliary disorders) | 1
Molluscum contagiosum (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neutropenic fever (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Non-cardiac chest pain (General disorders) | 1
Oral ulcer (General disorders) | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Pancytopenia (Investigations) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pharynx erythematous (General disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Right side flank pain (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Renal calculi (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinovirus (pos) (Infections and infestations) | 1
Shortness of breath (General disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Skin rash (Skin and subcutaneous tissue disorders) | 1
Sore throat (Infections and infestations) | 2
Subacute thyroiditis (Endocrine disorders) | 1
T-AML (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tachycardia (Cardiac disorders) | 1
Tender abdomen (General disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Weakness (General disorders) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02981914/Prot_SAP_000.pdf